CLINICAL TRIAL: NCT05974410
Title: Expanded Access to Immunomodulatory AVM0703 for Solid Tumor and Blood Cancer Patients
Status: Available | Type: Expanded Access
Sponsor: AVM Biotechnology Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: AVM0703-EAP
Record Dates: First submitted 2023-07-26; First posted 2023-08-03 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Glioblastoma; Squamous Cell Carcinoma; Hodgkin Lymphoma; Non-hodgkin Lymphoma; Breast Cancer; Prostate Cancer; Gastric Cancer; Ovarian Cancer; Acute Leukemia; Pancreatic Cancer; Spindle Cell Sarcoma; Cancer; Tumor, Solid; Tumor, Brain; Esophageal Andeocarcinoma; Mixed Phenotype AML; Desmoplastic Round Cell Sarcoma
MeSH Terms: conditions — Glioblastoma; Carcinoma, Squamous Cell; Hodgkin Disease; Lymphoma, Non-Hodgkin; Breast Neoplasms; Prostatic Neoplasms; Stomach Neoplasms; Ovarian Neoplasms; Pancreatic Neoplasms; Sarcoma; Neoplasms; Brain Neoplasms | interventions — Hydrocortisone; Proton Pump Inhibitors

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: AVM0703 — small molecule immunomodulatory drug
Drug: Hydrocortisone — physiologic circadian glucocorticoid
Drug: Proton pump inhibitor

SUMMARY:
AVM Biotechnology, Inc., provides immunomodulatory AVM0703 to solid tumor and blood cancer patients upon request by a US licensed MD or DO. As of July 2024, 37 patients have been treated through this FDA-EAP including patients diagnosed with relapsed or recurring glioblastoma, inoperable/chemotherapy ineligible CNS Squamous Cell Carcinoma, metastatic Breast Cancer, ovarian cancer, gastric cancer, Hodgkin's Lymphoma, Mixed Phenotype Acute Myelogenous Leukemia, colon cancer, B-ALL, Malignant Myxoid Spindle Cell Neoplasm, non-small cell lung cancer, DLBCL with CNS involvement, metastatic prostate cancer, Anaplastic T-cell Non-Hodgkin's Lymphoma and metastatic pancreatic cancer. Drug-related side-effects are predominantly grade 1 and include itching during the infusion and about 1 week of low grade insomnia.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Edward Loniewski, D.O., Study Director — AVM Biotechnology Inc